CLINICAL TRIAL: NCT00128635
Title: An Open-Label, Dose Confirmation and Dosimetry Study of Interstitial 131 I-chTNT-1/B MAb (COTARA(TM)) For the Treatment of Glioblastoma Multiforme (GBM) at 1st or 2nd Relapse
Brief Title: Iodine I 131 Monoclonal Antibody TNT-1/B in Treating Patients With Progressive or Recurrent Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000438768; NABTT-0404
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2007-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma; recurrent adult brain tumor
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — 131I-chimeric TNT-1-B monoclonal antibody

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody TNT-1/B

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies, such as iodine I 131 monoclonal antibody TNT-1/B (^131I MOAB TNT-1/B), can find tumor cells and carry tumor-killing substances to them without harming normal cells. This may be an effective treatment for glioblastoma multiforme.

PURPOSE: This phase I trial is studying the side effects and best dose of ^131I MOAB TNT-1/B in treating patients with progressive or recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of iodine I 131 monoclonal antibody TNT-1/B in patients with progressive or recurrent glioblastoma multiforme.

Secondary

* Determine the biodistribution and radiation dosimetry of this drug in these patients.
* Determine the toxicity and tolerability of this drug in these patients.
* Determine the overall survival, median time of survival, and 6-month survival of patients treated with this drug.

OUTLINE: This is an open-label, multicenter, dose-escalation study of therapeutic doses of iodine I 131 monoclonal antibody TNT-1/B (^131I MOAB TNT-1/B).

The first 12 patients accrued to the study undergo stereotactic placement of 2 catheters within the contrast-enhancing tumor on day 0. These patients then receive an imaging dose of ^131I MOAB TNT-1/B interstitially over approximately 25 hours on day 1 followed by dosimetry, biodistribution evaluations, and whole body imaging over an 8-10 day period. Beginning at least 2 weeks, but no more than 4 weeks later, all patients undergo catheter placement as above. One day later, patients receive a therapeutic dose of ^131I MOAB TNT-1/B interstitially over approximately 25 hours.

Cohorts of 3-6 patients receive escalating therapeutic doses of ^131I MOAB TNT-1/B until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 10 patients are treated at the MTD.

After completion of study treatment, patients are followed weekly for 3 weeks, at 6 weeks, at 4, 8, and 12 weeks (for the first 12 patients accrued to the study), every 4 weeks until disease progression, and then every 8 weeks thereafter.

PROJECTED ACCRUAL: Approximately 22 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme

  * Focal disease
  * Progressive or recurrent disease after prior treatment with radiotherapy and/or chemotherapy
  * Low-grade astrocytoma that progressed to glioblastoma multiforme after prior radiotherapy and/or chemotherapy allowed
* Gross tumor volume 5-60 mL
* No intraventricular tumor, infratentorial tumor, or tumor that communicates with the ventricles
* No bilateral non-contiguous gadolinium-enhancing tumor
* No diffuse disease, defined as any satellite lesion > 1.5 cm from the anticipated location of a catheter tip OR > 2 satellite lesions
* No ventricular invasion outside the anticipated radiotherapy volume

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9.0 g/dL

Hepatic

* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN)
* Hepatitis B negative
* No evidence of active hepatitis

Renal

* Creatinine ≤ 1.7 mg/dL
* BUN ≤ 2 times ULN

Cardiovascular

* No uncontrolled hypertension
* No unstable angina pectoris
* No uncontrolled cardiac dysrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to undergo MRI
* Mini Mental State Exam score ≥ 15
* No serious infection
* No other medical illness that would preclude study participation
* No other malignancy within the past 5 years except curatively treated carcinoma in situ or basal cell skin cancer
* No psychological or sociological condition, addictive disorder, or other condition that would preclude study compliance
* No known or suspected allergy to study drug or iodine
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior monoclonal antibodies
* No prior local immunotherapy or treatment with the following biologic agents:

  * Immunotoxins
  * Immunoconjugates
  * Antiangiogenesis compounds
  * Antisense agents
  * Peptide receptor antagonist
  * Interferons
  * Interleukins
  * Tumor infiltrating lymphocytes
  * Lymphokine-activated killer cells
  * Gene therapy

Chemotherapy

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* At least 3 months since prior polifeprosan 20 with carmustine implant (Gliadel wafer^® )

Endocrine therapy

* Must be maintained on a stable corticosteroid dose (approximately 4 mg) for ≥ 2 weeks before study entry

Radiotherapy

* See Disease Characteristics
* At least 3 months since prior radiotherapy
* No prior brachytherapy or radiosurgery

Surgery

* At least 4 weeks since prior surgery

Other

* Recovered from all prior therapy
* At least 1 month since prior investigational agents
* No more than 2 prior treatment regimens
* No other prior local therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2005-10; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose based on CTCAE v3.0 weekly for 8 weeks then every 8 weeks

SECONDARY OUTCOMES:
Biodistribution and radiation dosimetry by blood, urine, and whole body scans daily for 10 days
Toxicity by CTCAE v3.0 weekly for 12 weeks then every 8 weeks
Overall survival, median time of survival, and percent alive at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Lustig, MD, Study Chair — Abramson Cancer Center at Penn Medicine; Kevin Judy, MD — Abramson Cancer Center at Penn Medicine
Locations (4):
- United States (4):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama-Birmingham, Birmingham, Alabama
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania